CLINICAL TRIAL: NCT01981525
Title: A Pilot Study of Metformin in Patients With a Diagnosis of Li-Fraumeni Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140005; 14-C-0005
Record Dates: First submitted 2013-11-07; First posted 2013-11-11 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Li-Fraumeni Syndrome
Keywords: TP53 germline mutations
MeSH Terms: conditions — Li-Fraumeni Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Patients will receive metformin at level 1 dose for 2 weeks. If dose is tolerated, patient will receive level 2 dose for 2 weeks and if tolerated will escalate to level 3 dose, and if tolerated will escalate to level 4 dose.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Treatment will be administered primarily on an outpatient basis. Patients will be instructed to take 500 mg metformin by mouth 1, 2 or 3 times a day or 1000 mg twice per day depending on dose level. Patients will receive metformin at level 1 dose for 2 weeks. If dose is tolerated, patient will receive level 2 dose for 2 weeks and if tolerated will escalate to level 3 dose, and if tolerated will escalate to level 4 dose. Metformin will be taken for 14 weeks.

SUMMARY:
Background:

* Li Fraumeni Syndrome (LFS) is a highly penetrant, autosomal dominant cancer predisposition disorder. Four main cancer types including sarcoma, adrenocortical carcinoma, breast cancer, and malignant brain tumors commonly characterize LFS but the syndrome can include other cancers.
* Metformin is an oral biguanide drug that is approved by the FDA for the treatment of type II diabetes. Metformin has been associated with reduced cancer risk in several epidemiologic studies and reduced cancer mortality in patients with type 2 diabetes.
* Metformin decreases circulating insulin and IGF1, and promotes glucose uptake in skeletal muscle and inhibits gluconeogenesis in the liver. Elevations in circulating insulin and IGF1 levels have been associated with increased cancer risk.
* Preclinical research in animal models shows that metformin may be more toxic in cancer cells that have lost p53 function.
* Lifetime risk of cancer in LFS patients with germline TP53 mutations is estimated to be up to 70% by age 60, with women having excess lifetime cancer risk (up to 100%) compared to men (up to 80%). There are currently no approved chemopreventive agents for patients with LFS.
* Metformin has been shown to be safe and tolerable in diabetic and non-diabetics, and may be an ideal candidate for chemoprevention of cancer in this population.

Objectives:

* Determine the tolerability of oral daily metformin in patients with LFS caused by germline TP53 mutations.
* Determine if 8 weeks of daily metformin administration has any effect on circulating IGF-1, insulin, and IGFBP3

Eligibility:

* Must have a germline TP53 mutation and provide documentation of testing.
* Must have adequate organ function.
* Age greater than or equal to 18 years.

Design:

* This is a pilot study to assess the tolerability of daily oral metformin administration in patients with LFS caused by germline TP53 mutations and to study the effect of metformin on biomarker levels in these subjects.
* In the absence of intolerable toxicity, a minimum of 22 patients will take metformin by mouth for a total of 14 weeks and then discontinue metformin for 6 weeks. The total time on study will be 20 weeks.
* Patients will be assessed for biomarker levels (IGF-1, insulin, IGFBP3) by blood sample at baseline, and weeks 0 and 8.

DETAILED DESCRIPTION:
Background:

* Li Fraumeni Syndrome (LFS) is a highly penetrant, autosomal dominant cancer predisposition disorder. Four main cancer types including sarcoma, adrenocortical carcinoma, breast cancer, and malignant brain tumors commonly characterize LFS but the syndrome can include other cancers.
* Metformin is an oral biguanide drug that is approved by the FDA for the treatment of type II diabetes. Metformin has been associated with reduced cancer risk in several epidemiologic studies and reduced cancer mortality in patients with type 2 diabetes.
* Metformin decreases circulating insulin and IGF1, and promotes glucose uptake in skeletal muscle and inhibits gluconeogenesis in the liver. Elevations in circulating insulin and IGF1 levels have been associated with increased cancer risk.
* Preclinical research in animal models shows that metformin may be more toxic in cancer cells that have lost p53 function.
* Lifetime risk of cancer in LFS patients with germline TP53 mutations is estimated to be up to 70% by age 60, with women having excess lifetime cancer risk (up to 100%) compared to men (up to 80%). There are currently no approved chemopreventive agents for patients with LFS.
* Metformin has been shown to be safe and tolerable in diabetic and non-diabetics, and may be an ideal candidate for chemoprevention of cancer in this population.

Objectives:

* Determine the tolerability of oral daily metformin in patients with LFS caused by germline TP53 mutations.
* Determine if 8 weeks of daily metformin administration has any effect on circulating IGF-1, insulin, and IGFBP3

Eligibility:

* Must have a germline TP53 mutation and provide documentation of testing.
* Must have adequate organ function.
* Age greater than or equal to 18 years.

Design:

* This is a pilot study to assess the tolerability of daily oral metformin administration in patients with LFS caused by germline TP53 mutations and to study the effect of metformin on biomarker levels in these subjects.
* In the absence of intolerable toxicity, a minimum of 22 patients will take metformin by mouth for a total of 14 weeks and then discontinue metformin for 6 weeks. The total time on study will be 20 weeks.
* Patients will be assessed for biomarker levels (IGF-1, insulin, IGFBP3) by blood sample at baseline, and weeks 0, 8, 14 and 20.

ELIGIBILITY:
* INCLUSION CRITERIA:
* All TP53 germline mutation positive adult patients will be eligible for this study. All patients must have a documented TP53 germline mutation.
* Patients with history of cancer must be in remission, with surgery completed at least 6 months prior to enrollment and chemotherapy completed at least 1 year prior to enrollment (except for basel cell carcinoma of the skin).
* Age greater than or equal to 18 years. The doses of metformin used in this study exceed the maximum recommended daily dose for the pediatric population.
* ECOG performance status 0 or 1 or Karnofsky greater than or equal to 70%
* Patients must have normal organ and marrow function as defined below:

  * Leukocytes*: greater than or equal to 3,000/microL*
  * Absolute neutrophil count: greater than or equal to 1,500/ microL
  * Platelets: greater than or equal to 100,000/ microL
  * Total bilirubin: Within normal institutional limits
  * AST(SGOT) / ALT(SGPT): less than or equal to 2.5 times institutional upper limit of normal
  * Creatinine: Within normal institutional limits OR
  * Creatinine clearance: greater than or equal to 60 mL/min/1.73m(2) if serum creatinine > institutional normal

    * Note: If leukopenia is idiopathic and no other significant co-morbidities exist patients will not be excluded on the basis of their WBC.
* Metformin is a category B drug and can be used to treat gestational diabetes. Levels of metformin excreted in breast milk appear to be low and not clinically significant. However, for protocol safety reasons, we will not be enrolling pregnant and/or nursing women in this study as metformin as has not been extensively evaluated in non-diabetic pregnant and nursing women. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Women who are nursing will be advised to discontinue breastfeeding if the mother is treated with metformin. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform Drs. Annunziata or Walcott, or protocol physicians/study team at NCI and her primary care provider immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document.

GENERAL EXCLUSION CRITERIA:

* Patients who have had stem-cell transplantation.
* Current use of metformin or other anti-diabetic agents, or hypersensitivity or allergy to metformin.
* Patients who are receiving any other investigational agents.
* Patients with history of chronic alcohol use
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin or other agents used in study.
* Patients with congestive heart failure requiring pharmacological management.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

EXCLUSION CRITERIA for 13C-MBT STUDIES:

Exclusion criteria for 13C-MBT studies in addition to general exclusion criteria (pertaining to effects of oral uptake of the administered substrate or mitochondrial function in the liver):

* Gastric paresis
* Short gut syndrome
* Inflammatory bowel disease*
* Celiac sprue
* Pancreatic insufficiency or disease
* Any malabsorption disease/syndrome
* Chronic PPI use or H2 blocker use that cannot be temporarily discontinued (at least 48 hours)
* Any acetaminophen, aspirin, NSAID, or statin use within 2 days of testing (known to affect mitochondrial function)
* Drugs that interfere with mitochondrial function if they are unable to be discontinued 48 hours prior to (13)MBT testing will be excluded for this test only but eligible for the rest of the protocol.
* Any oral steroid use within 2 weeks of testing
* Chronic alcohol use** defined as > 2 standard drinks per day (more than 2 beers, 2 glasses of wine, or 2 shots of liquor per day)

  * Inflammatory bowel disease will be exclusion for the (13)C-MBT only, because even if well controlled we do not know the effect chronic inflammation in the bowel and steroid use may have on the test. The test analyzes exhaled CO2 in the breath and this can be affected by diet (carbohydrate heavy), exercise, and certain pathologies like liver disease. Also pro-inflammatory mediators have been shown to cause hepatocellular injury that may also interfere with results of the test.

    * The test is currently being studied as an early detection, non-invasive method for liver cirrhosis. Therefore, patients who have had chronic alcohol use consistent with a regular pattern of alcohol consumption may have underlying liver disease that may affect the CO2 measurement. Further, alcohol changes the NADH/NAD ratio intracellularly and studies have shown that alcohol can inhibit methionine oxidation. Previous protocols utilizing the (13)C-MBT have excluded patients who consume greater than 20 g/day of alcohol. A standard drink is equivalent to approximately 14 g/day of alcohol (one 12 oz beer, one 5 oz glass of wine, or one shot of liquor). This information was obtained from the National Institute of Health/National Institute of Alcohol Abuse and Alcoholism (NIAAA):

http://pubs.niaaa.nih.gov/publications/Practitioner/pocketguide/pocket_guide2.htm). We will also evaluate LFTs and should clinical concern arise, check PT/PTT and albumin. Patients with normal liver function and no substantial history of alcohol abuse will be eligible.

EXCLUSION CRITERIA FOR 31P-MRS STUDIES:

Although patients will need to sign a separate informed consent to undergo the (31)P-MRS studies the list below includes some of the general exclusion criteria as information for the caring physician. Exclusion criteria for (31)P-MRS studies in addition to general exclusion criteria:

* Inability to perform exercise with dominant leg
* Claustrophobia and/or inability to lie flat in MRI machine
* Metal medical implantable device or other MRI incompatible materials
* Body mass index under 19 or over 45
* Prior stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-01-27 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Determine the tolerability of metformin in patients with LFS caused by germline TP53 mutations | 2 years
  toxicity assessment by CTCAE ver 4.0
Determine if 8 weeks of daily metformin administration has any effect on circulating IGF-1, insulin, and IGFBP3 | 2 years
  biomarker levels (IGF-1, insulin, IGFBP3) by blood sample at baseline, and weeks 0, 8, 14 and 20

SECONDARY OUTCOMES:
Determine if daily metformin administration has any effect on circulating IGF-1, insulin, and IGFBP3 levels, two weeks after the start of metformin administration and six weeks after discontinuing metformin (week 20) | 2 years
  toxicity classification by NCI Common Terminology Criteria for Adverse Events (CTCAE)
Determine if daily metformin administration has any effect on skeletalmuscle mitochondrial function using phosphorous-31 magnetic resonance spectroscopy (31P-MRS) baseline and eight weeks after the start of metformin. | 2 years
  biomarker levels (IGF-1, insulin, IGFBP3) by blood sample at baseline, and weeks 0, 8, 14 and 20

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Annunziata, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Li FP, Fraumeni JF Jr. Soft-tissue sarcomas, breast cancer, and other neoplasms. A familial syndrome? Ann Intern Med. 1969 Oct;71(4):747-52. doi: 10.7326/0003-4819-71-4-747. No abstract available. PMID 5360287
- [Background] Li FP, Fraumeni JF Jr, Mulvihill JJ, Blattner WA, Dreyfus MG, Tucker MA, Miller RW. A cancer family syndrome in twenty-four kindreds. Cancer Res. 1988 Sep 15;48(18):5358-62. PMID 3409256
- [Background] Villani A, Tabori U, Schiffman J, Shlien A, Beyene J, Druker H, Novokmet A, Finlay J, Malkin D. Biochemical and imaging surveillance in germline TP53 mutation carriers with Li-Fraumeni syndrome: a prospective observational study. Lancet Oncol. 2011 Jun;12(6):559-67. doi: 10.1016/S1470-2045(11)70119-X. Epub 2011 May 19. PMID 21601526
- [Derived] Wang PY, Li J, Walcott FL, Kang JG, Starost MF, Talagala SL, Zhuang J, Park JH, Huffstutler RD, Bryla CM, Mai PL, Pollak M, Annunziata CM, Savage SA, Fojo AT, Hwang PM. Inhibiting mitochondrial respiration prevents cancer in a mouse model of Li-Fraumeni syndrome. J Clin Invest. 2017 Jan 3;127(1):132-136. doi: 10.1172/JCI88668. Epub 2016 Nov 21. PMID 27869650
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0005.html